CLINICAL TRIAL: NCT01712464
Title: Modulation of Reinforcement Learning and Neuronal Activation in Ventral Stratum by Oxytocin - a Pilot Study at Autism Spectrum Disorder
Brief Title: Modulation of Reinforcement Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 12-033
Record Dates: First submitted 2012-10-15; First posted 2012-10-23 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Impact of Oxytocin on Social Learning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cross over Oxytocin and Placebo (Other): FMRI measurement and blood examinations after 26 IU Oxytocin (Syntocinon)or placebo on two consecutive days
  Interventions: Drug: Oxytocin vs. Placebo
- Cross over Placebo and Oxytocin (Other): FMRI measurement and blood examinations after 26 IU Oxytocin (Syntocinon)or placebo on two consecutive days
  Interventions: Drug: Oxytocin vs. Placebo

INTERVENTIONS:
Drug: Oxytocin vs. Placebo — FMRI measurement and blood examinations after 26 IU Oxytocin (Syntocinon)or placebo on two consecutive days

SUMMARY:
This study aims to examine the modulation of neuronal and behavioural parameters of social reinforcement learning.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 26 years
* male
* IQ>80
* written informed consent
* proband understands character, extent and individual consequences of the study
* competent persons who are able to follow the instructions of the study personnel
* for ASD patients: assured ASD diagnosis, comply of the ASD criteria ADI-R/ADOS-G

Exclusion Criteria:

* prosopagnosia
* anaphylaxis of oxytocin or other chemical substances
* metal inside the body or other contraindications of mri scan
* physical illness which can affect the examinations or endanger the proband
* actual or assumed drug or alcohol abuse
* persons who are accommodated in an institution because of court or administrative order
* persons with a relationship of dependence to the sponsor or investigator
* healthy probands: psychiatric disorder according to ICD-10-WHO F at the moment and in history, continuous drug-intake at time of measurements
* patients with ASD: psychiatric disorder according to ICD-10-WHO F (except ASD disorder in patient group) during the last 12 month being not treated, continuous drug-intake at time of measurements (psychotropic medication), exception: stimulants used for treatment of attention disorders, if they can come off for the measurements

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2016-08-07 (Actual); Study Completion 2016-08-07 (Actual)

PRIMARY OUTCOMES:
Bold Signal in nucleus accumbens | 1 Day
  during social learning at one treatment with oxytocin vs placebo

SECONDARY OUTCOMES:
Bold signal in ventral tegmental areal | 1 Day
  during social learning at one treatment with oxytocin vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schulte-Rüther, Dr. rer. nat, Study Director — University Hospital, Aachen
Locations (1):
- Universtiy Hospital Aachen, Aachen, Northrhine-Westfalia, Germany